CLINICAL TRIAL: NCT00450684
Title: Cardiac Resynchronization Therapy in Heart Failure Patients With Congenital Heart Defects
Brief Title: Cardiac Resynchronization Therapy in Congenital Heart Defects
Acronym: CARE-CHD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARE-CHD
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group A (Experimental): Implantation and testing of CRT
  Interventions: Device: Implantation and testing of CRT
- Group B (Experimental): IImplantation and testing of CRT
  Interventions: Device: Implantation and testing of CRT

INTERVENTIONS:
Device: Implantation and testing of CRT — Biventricular pacing for 12 weeks (CRT ON) followed by automatic rhythmicity or the original, conventional biventricular stimulation for 12 weeks (CRT OFF), then returning to biventricular pacing (CRT ON).
Device: Implantation and testing of CRT — Automatic rhythmicity or original conventional biventricular stimulation for 12 weeks (CRT OFF) followed by biventricular pacing (CRT ON).

SUMMARY:
The objective of this multicentre prospective therapeutic study is to evaluate the effects of CRT on the right and left ventricular function of patients with CHD in the medium and long term. Patients who reject the randomization or cannot be paced with right ventricular pacing alone will be enrolled in group C with continuous biventricular pacing, which is the main group in this study. Optional: Immediately after implantation the patients are divided into group A and B (randomized, single blind (for the patient), cross-over design).

The treatment and the completing follow-up examination will take approximately 18 months and includes seven visits - one previous to the CRT and six at certain times afterward. At selected time intervals echocardiographic 3D and Tissue Doppler Imaging to evaluate the global and regional ventricular function are performed. Subjective quality of life assessment (questionnaire) will also be performed at the defined follow-up intervals, and if applicable (optional) also objective assessment of the physical performance (VO2 max).

55 patients also including children and adults with CHD are planned to be included in the study. The main target is to provide evidence of the effectiveness of CRT with biventricular stimulation in terms of improved ventricular function (ejection fraction and QRS interval).

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart defects
* Heart failure of the Morphologically right or left system ventricle with an absolute ejection fraction of < 40% in the failed ventricle
* NYHA classes II-IV
* Optimal drug therapy for heart failure according to the ESC guidelines
* QRS interval ≥ 120 ms (demonstrated in at least two relevant ECG derivations, depending on existing bundle branch block symptoms)
* Patients with chronic stimulation of the subpulmonary ventricle by a 1- or 2-ventricle pacemaker, which also meets the above-mentioned criteria
* Patients with morphologically right ventricle in system position and significant insufficiency of the systemic atrioventricular valve, if they also meet the criteria listed above

Exclusion Criteria:

* PTCA, cardiomyoplasty or myocardial infarction / unstable angina pectoris or cerebral insult within the 6 weeks preceding the planned cardiac resynchronisation therapy
* Patients with pulmonary hypertension / Eisenmenger's syndrome
* Life expectancy < 1 year due to a non-cardiac disease
* Anticipated poor compliance by the patient
* Pregnancy and breastfeeding
* Known or persistent abuse of prescription medicines, recreational drugs or alcohol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 7 visits
QRS-interval | 7 visits

SECONDARY OUTCOMES:
Echocardiographic standard parameters (e.g. LVIDd. FS, RVIDd) | 7 visits
Tissue Doppler echocardiography: dyssynchrony parameters, regional myocardiac function | 7 visits
3D echocardiography:LV volumes, LVEF, Dyssynchrony index | 7 visits
NT pro-BNP | 7 visits
Spiroergometry: performance P (W/kg), incl. VO2,max | 6 visits
Walking distance in 6 minutes | 6 visits
Decrease of hospitalization | 18 months
Decrease of ventricular and atrial arrhythmias | 18 months
Prevention or postponement of heart transplantation | 18 Months
Quality of life | 6 visits
death | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Abdul-Khaliq, Prof., MD, Principal Investigator — Competence Network for Congenital Heart Defects
Locations (16):
- AKH Wien, Klinische Abteilung für Pädiatrische Kardiologie, Vienna, Austria
- Germany (15):
  - Universitätsklinikum Münster, Klinik für angeborene (EMAH) und erworbene Herzfehler, Münster, North Rhine-Westphalia
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Pädiatrische Kardiologie, Halle, Saxony-Anhalt
  - Uniklinik RWTH Aachen, AÖR, Klinik für Kinderkardiologie, Aachen
  - Herz- und Diabeteszentrum NRW, Klinik für Kinderkardiologie und angeborene Herzfehler, Bad Oeynhausen
  - Charité - Universitätsmedizin Berlin, Klinik für Pädiatrie mit Schwerpunkt Kardiologie, Berlin
  - Deutsches Herzzentrum Berlin, Klinik für Angeborene Herzfehler/Kinderkardiologie, Berlin
  - Elektrophysiologie Bremen und Herzzentrum Bremen, Abteilung für Angeborene Herzfehler/Kinderkardiologie, Bremen
  - Universitätsklinikum Erlangen, Kinderkardiologische Abteilung, Erlangen
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Zentrum für Kinder- und Jugendmedizin, Angeborene Herzfehler/Pädiatrische Kardiologie, Freiburg im Breisgau
  - Universitäres Herzzentrum Hamburg, Kinderkardiologie, Hamburg
  - Universitätsklinikum des Saarlandes, Klinik für Pädiatrische Kardiologie, Homburg/Saar
  - Deutsches Herzzentrum München, Klinik für Kinderkardiologie und angeborene Herzfehler, München
  - Universitätsklinikum Münster, Klinik und Poliklinik für Kinder- und Jugendmedizin, Pädiatrische Kardiologie, Münster
  - Deutsches Kinderherzzentrum Sankt Augustin, Abt. Kardiologie/Angeborene Herzfehler, Sankt Augustin
  - Universitätsklinik für Kinder- und Jugendmedizin Tübingen, Abt. Kinderkardiologie, Pulmologie, Intensivmedizin, Tübingen

REFERENCES:
- See also: Related Info — http://www.kompetenznetz-ahf.de